CLINICAL TRIAL: NCT01486290
Title: Identifying and Overcoming Barriers to Diabetes Management in the Elderly: A Cost-effective Intervention Study
Acronym: DISCO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joslin Diabetes Center (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Principal Investigator, Medha Munshi, Director of Geriactric Diabetes Clinic, Joslin Diabetes Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 07-03
Record Dates: First submitted 2011-11-23; First posted 2011-12-06 (Estimated); Last update posted 2014-03-28 (Estimated); Status verified 2014-03

CONDITIONS: Diabetes
Keywords: Intervention; Cost Effective; Elderly; Glycemic Control
MeSH Terms: conditions — Diabetes Mellitus | interventions — Educational Status; Nutritional Status

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Geriatric Diabetes Team Intervention (Experimental): The subjects in this group underwent evaluation for barriers to self care by a diabetes educator well versed with age specific barriers. After consideration of patient clinical, function, and psychosocial background, a geriatric diabetes team devised strategy to help patients cope with respective barriers. An office based diabetes diabetes educator conveyed the strategy to patient and caregivers viz phone calls. the educator called study participants up wot eleven times over a sex month period.
  Interventions: Behavioral: Behavioral
- Atention Control Arm (No Intervention): The subjects in the group received similar, in person contact, as the intervention group. an educator, separate from the one involved in the intervention team, called patients in this group for a total of eleven times within the first six months. The Phone calls were focused toward general discussion without any diabetes related advice.

INTERVENTIONS:
Behavioral: Behavioral — the intervention included developing strategies to help patients cope with their barriers to self care. The intervention were implemented by an office based educator over a six month by phone calls. From six months to twelve months subjects did not have any contact with study staff.
  Other Names: Clinical; Education; Nutrition; Care coordination
  Arms: Geriatric Diabetes Team Intervention

SUMMARY:
The purpose of this study is to find ways to identify barriers that affect self care in older adult with diabetes and to provide cost effective coping strategies to improve clinical, functional and psychosocial measures.

DETAILED DESCRIPTION:
This is a study to evaluate whether short term focused intervention by a geriatric diabetes team to help overcome barriers to diabetes care in older adults will result in improved clinical, functional, and quality of life measures compared to usual care in a cost effective manner. In addition, we will assess whether the support network formed during intervention by the geriatric diabetes team will empower patients, resulting in long lasting improvement in parameters after intervention is completed.

ELIGIBILITY:
Inclusion Criteria:

* Age 70 years and older
* Diagnosis of type 1 or type 2 diabetes
* Seen at Joslin Clinic or Beth Israel Deaconess Medical Center for at least one year
* HbA1c 8% X 2 in past 6 months without fluctuation of more than 0.5% (i.e. stable poor control)
* No major change in medications in past 3 months, e.g. addition of insulin or another hypoglycemic agent

Exclusion Criteria:

* Patients with terminal diseases, e.g. malignancy with expected life expectancy of 12 months or less
* Patients who live more than 25 miles from Joslin Clinic/Beth Israel Deaconess Medical Center
* Patients who live in an institutional setting (e.g. nursing home, group home, etc)
* Patients who are not able to complete outcome assessments, (e.g. poor vision, diminished mental capacity/severe cognitive decline, unable to speak/read/write English

Min Age: 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 52 (Actual)
Dates: Start 2007-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1c | 6 and 12 months
  The primary outcomes of the study is to measure change in A1c before and after intervention.

SECONDARY OUTCOMES:
Hypoglycemia | 6 and 12 months
  Frequency of hypoglycemia by history and by hypoglycemia calendar
functionality | 6 and 12 months
  6-minute walk test, Tinetti test, number of falls and fear of falls, activities of daily living and instrumental activities of daily living
Cognitive function | 6 and 12 months
  cognitive function test by modified clock drawing test, verbal fluency and Trail-making tests A and B
Depression | 6 and 12 months
  Geriatric depression scale
Self care inventory - revised | 6 and 12 months
  frequency of self-care measures
Problem areas in diabetes | 6 and 12 months
  Measure of diabetes-related distress
Economic impact | 6 and 12 months
  number of emergency room visit, hospitalizations for diabetes-related illnesses, out-patient care utilization in the form of clinic visits

CONTACTS AND LOCATIONS:
Overall Officials: Medha N Munshi, MD, Principal Investigator — Joslin Diabetes Center
Locations (1):
- Joslin Diabetes Center, Boston, Massachusetts, United States

REFERENCES:
- [Background] Makimattila S, Malmberg-Ceder K, Hakkinen AM, Vuori K, Salonen O, Summanen P, Yki-Jarvinen H, Kaste M, Heikkinen S, Lundbom N, Roine RO. Brain metabolic alterations in patients with type 1 diabetes-hyperglycemia-induced injury. J Cereb Blood Flow Metab. 2004 Dec;24(12):1393-9. doi: 10.1097/01.WCB.0000143700.15489.B2. PMID 15625413
- [Background] Norris SL, Nichols PJ, Caspersen CJ, Glasgow RE, Engelgau MM, Jack L, Isham G, Snyder SR, Carande-Kulis VG, Garfield S, Briss P, McCulloch D. The effectiveness of disease and case management for people with diabetes. A systematic review. Am J Prev Med. 2002 May;22(4 Suppl):15-38. doi: 10.1016/s0749-3797(02)00423-3. PMID 11985933
- [Background] Fordyce M, Bardole D, Romer L, Soghikian K, Fireman B. Senior Team Assessment and Referral Program--STAR. J Am Board Fam Pract. 1997 Nov-Dec;10(6):398-406. PMID 9407480
- [Background] Munshi M, Grande L, Hayes M, Ayres D, Suhl E, Capelson R, Lin S, Milberg W, Weinger K. Cognitive dysfunction is associated with poor diabetes control in older adults. Diabetes Care. 2006 Aug;29(8):1794-9. doi: 10.2337/dc06-0506. PMID 16873782
- [Background] Blaum CS, Ofstedal MB, Langa KM, Wray LA. Functional status and health outcomes in older americans with diabetes mellitus. J Am Geriatr Soc. 2003 Jun;51(6):745-53. doi: 10.1046/j.1365-2389.2003.51256.x. PMID 12757559
- [Background] Bertoni AG, Kirk JK, Goff DC Jr, Wagenknecht LE. Excess mortality related to diabetes mellitus in elderly Medicare beneficiaries. Ann Epidemiol. 2004 May;14(5):362-7. doi: 10.1016/j.annepidem.2003.09.004. PMID 15177276
- [Background] Economic consequences of diabetes mellitus in the U.S. in 1997. American Diabetes Association. Diabetes Care. 1998 Feb;21(2):296-309. doi: 10.2337/diacare.21.2.296. PMID 9539999
- [Background] Brown AF, Mangione CM, Saliba D, Sarkisian CA; California Healthcare Foundation/American Geriatrics Society Panel on Improving Care for Elders with Diabetes. Guidelines for improving the care of the older person with diabetes mellitus. J Am Geriatr Soc. 2003 May;51(5 Suppl Guidelines):S265-80. doi: 10.1046/j.1532-5415.51.5s.1.x. No abstract available. PMID 12694461
- [Background] Task Force on Community Preventive Services. Recommendations for healthcare system and self-management education interventions to reduce morbidity and mortality from diabetes. Am J Prev Med. 2002 May;22(4 Suppl):10-4. doi: 10.1016/s0749-3797(02)00422-1. No abstract available. PMID 11985932
- [Background] Baird TA, Parsons MW, Barber PA, Butcher KS, Desmond PM, Tress BM, Colman PG, Jerums G, Chambers BR, Davis SM. The influence of diabetes mellitus and hyperglycaemia on stroke incidence and outcome. J Clin Neurosci. 2002 Nov;9(6):618-26. doi: 10.1054/jocn.2002.1081. PMID 12604269
- [Background] Fulesdi B, Limburg M, Bereczki D, Kaplar M, Molnar C, Kappelmayer J, Neuwirth G, Csiba L. Cerebrovascular reactivity and reserve capacity in type II diabetes mellitus. J Diabetes Complications. 1999 Jul-Aug;13(4):191-9. doi: 10.1016/s1056-8727(99)00044-6. PMID 10616858
- [Background] Griffith DN, Saimbi S, Lewis C, Tolfree S, Betteridge DJ. Abnormal cerebrovascular carbon dioxide reactivity in people with diabetes. Diabet Med. 1987 May-Jun;4(3):217-20. doi: 10.1111/j.1464-5491.1987.tb00865.x. PMID 2956022
- [Background] Kadoi Y, Hinohara H, Kunimoto F, Saito S, Ide M, Hiraoka H, Kawahara F, Goto F. Diabetic patients have an impaired cerebral vasodilatory response to hypercapnia under propofol anesthesia. Stroke. 2003 Oct;34(10):2399-403. doi: 10.1161/01.STR.0000090471.28672.65. Epub 2003 Sep 4. PMID 12958324
- [Background] Jimenez-Bonilla JF, Carril JM, Quirce R, Gomez-Barquin R, Amado JA, Gutierrez-Mendiguchia C. Assessment of cerebral blood flow in diabetic patients with no clinical history of neurological disease. Nucl Med Commun. 1996 Sep;17(9):790-4. doi: 10.1097/00006231-199609000-00009. PMID 8895906
- [Background] MacLeod KM, Gold AE, Ebmeier KP, Hepburn DA, Deary IJ, Goodwin GM, Frier BM. The effects of acute hypoglycemia on relative cerebral blood flow distribution in patients with type I (insulin-dependent) diabetes and impaired hypoglycemia awareness. Metabolism. 1996 Aug;45(8):974-80. doi: 10.1016/s0026-0495(96)90266-8. PMID 8769355
- [Background] KATZ S, FORD AB, MOSKOWITZ RW, JACKSON BA, JAFFE MW. STUDIES OF ILLNESS IN THE AGED. THE INDEX OF ADL: A STANDARDIZED MEASURE OF BIOLOGICAL AND PSYCHOSOCIAL FUNCTION. JAMA. 1963 Sep 21;185:914-9. doi: 10.1001/jama.1963.03060120024016. No abstract available. PMID 14044222
- [Background] Bean JF, Kiely DK, Leveille SG, Herman S, Huynh C, Fielding R, Frontera W. The 6-minute walk test in mobility-limited elders: what is being measured? J Gerontol A Biol Sci Med Sci. 2002 Nov;57(11):M751-6. doi: 10.1093/gerona/57.11.m751. PMID 12403805
- [Background] Lord SR, Menz HB. Physiologic, psychologic, and health predictors of 6-minute walk performance in older people. Arch Phys Med Rehabil. 2002 Jul;83(7):907-11. doi: 10.1053/apmr.2002.33227. PMID 12098148
- [Background] Bautmans I, Lambert M, Mets T. The six-minute walk test in community dwelling elderly: influence of health status. BMC Geriatr. 2004 Jul 23;4:6. doi: 10.1186/1471-2318-4-6. PMID 15272934
- [Background] Montorio I, Izal M. The Geriatric Depression Scale: a review of its development and utility. Int Psychogeriatr. 1996 Spring;8(1):103-12. doi: 10.1017/s1041610296002505. PMID 8805091
- [Background] Welch G, Weinger K, Anderson B, Polonsky WH. Responsiveness of the Problem Areas In Diabetes (PAID) questionnaire. Diabet Med. 2003 Jan;20(1):69-72. doi: 10.1046/j.1464-5491.2003.00832.x. PMID 12519323
- [Background] Tiecks FP, Lam AM, Aaslid R, Newell DW. Comparison of static and dynamic cerebral autoregulation measurements. Stroke. 1995 Jun;26(6):1014-9. doi: 10.1161/01.str.26.6.1014. PMID 7762016
- [Background] Panerai RB. Assessment of cerebral pressure autoregulation in humans--a review of measurement methods. Physiol Meas. 1998 Aug;19(3):305-38. doi: 10.1088/0967-3334/19/3/001. PMID 9735883
- [Background] Aaslid R, Newell DW, Stooss R, Sorteberg W, Lindegaard KF. Assessment of cerebral autoregulation dynamics from simultaneous arterial and venous transcranial Doppler recordings in humans. Stroke. 1991 Sep;22(9):1148-54. doi: 10.1161/01.str.22.9.1148. PMID 1926257
- [Background] Zhang R, Zuckerman JH, Giller CA, Levine BD. Transfer function analysis of dynamic cerebral autoregulation in humans. Am J Physiol. 1998 Jan;274(1 Pt 2):H233-41. doi: 10.1152/ajpheart.1998.274.1.h233. PMID 9458872
- [Background] Panerai RB, Dawson SL, Potter JF. Linear and nonlinear analysis of human dynamic cerebral autoregulation. Am J Physiol. 1999 Sep;277(3):H1089-99. doi: 10.1152/ajpheart.1999.277.3.H1089. PMID 10484432
- [Background] Lipsitz LA, Mukai S, Hamner J, Gagnon M, Babikian V. Dynamic regulation of middle cerebral artery blood flow velocity in aging and hypertension. Stroke. 2000 Aug;31(8):1897-903. doi: 10.1161/01.str.31.8.1897. PMID 10926954
- [Background] Benarroch EE, S.P., Low PA, The Valsalva Manuever. In Clinical Autonomic Disroders: Evaluation and Management, L.P. editor, Editor. 1993, Little Brown and company: Boston. p. 209-215.
- [Background] Rutan GH, Hermanson B, Bild DE, Kittner SJ, LaBaw F, Tell GS. Orthostatic hypotension in older adults. The Cardiovascular Health Study. CHS Collaborative Research Group. Hypertension. 1992 Jun;19(6 Pt 1):508-19. doi: 10.1161/01.hyp.19.6.508. PMID 1592445
- [Background] Low, P.A., Laboratory Evaluation of Autonomic Function. In Clinical Autonomic Disorders, P.A. Low, Editor. 1997, LIppincott-Raven: Philadelphia. p. 179-208.
- [Background] Novak V, Chowdhary A, Farrar B, Nagaraja H, Braun J, Kanard R, Novak P, Slivka A. Altered cerebral vasoregulation in hypertension and stroke. Neurology. 2003 May 27;60(10):1657-63. doi: 10.1212/01.wnl.0000068023.14587.06. PMID 12771258
- [Background] Greenfield JC Jr, Rembert JC, Tindall GT. Transient changes in cerebral vascular resistance during the Valsalva maneuver in man. Stroke. 1984 Jan-Feb;15(1):76-9. doi: 10.1161/01.str.15.1.76. PMID 6229907
- [Background] Werner C, Kochs E, Hoffman WE, Blanc IF, Schulte am Esch J. Cerebral blood flow and cerebral blood flow velocity during angiotensin-induced arterial hypertension in dogs. Can J Anaesth. 1993 Aug;40(8):755-60. doi: 10.1007/BF03009772. PMID 8403159
- [Derived] Munshi MN, Segal AR, Suhl E, Ryan C, Sternthal A, Giusti J, Lee Y, Fitzgerald S, Staum E, Bonsignor P, DesRochers L, McCartney R, Weinger K. Assessment of barriers to improve diabetes management in older adults: a randomized controlled study. Diabetes Care. 2013 Mar;36(3):543-9. doi: 10.2337/dc12-1303. Epub 2012 Nov 27. PMID 23193208